CLINICAL TRIAL: NCT07280910
Title: Retrospective Observational Study Analyzing De-identified Data Originally Collected as Part of a Quality Improvement (QI) Initiative.
Brief Title: Exploring Virtual Reality in Clinical Care - Impacts on Patient Distress, Parental Anxiety and Nurse Satisfaction
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20032312
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Anxiety
Keywords: Virtual Reality; Quality Improvement; Protected Health Information; Heart Rate; Blood Pressure; State-Trait Anxiety Inventory
MeSH Terms: conditions — Anxiety Disorders | interventions — Nurses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pediatric Patients: Pediatric patients receiving VR interventions (6-15 years)
  Interventions: Other: Virtual Reality
- Parent Caregivers: Parents of Pediatric patients receiving VR interventions (6-15 years)
  Interventions: Behavioral: Survey Responses/Parent Caregivers
- Nurses: The nursing staff are involved in the care process of the Pediatric patients receiving VR interventions (6-15 years)
  Interventions: Behavioral: Survey Responses/Nurses

INTERVENTIONS:
Other: Virtual Reality — Administered as part of a QI initiative aimed at reducing anxiety in pediatric patients during clinical care. The intervention involved using a VR system to provide a distraction and relaxation tool during routine procedures. This approach is consistent with recent research showing that VR can be an effective tool for reducing pain and anxiety in pediatric patients undergoing medical procedures. Retrospective data collection.
  Groups: Pediatric Patients
Behavioral: Survey Responses/Parent Caregivers — Survey responses from parents regarding anxiety and satisfaction.
  Groups: Parent Caregivers
Behavioral: Survey Responses/Nurses — Survey responses from nurses regarding anxiety and satisfaction.
  Groups: Nurses

SUMMARY:
Prior experience with virtual reality (VR) in clinical care has demonstrated its potential to reduce patient anxiety and distress, particularly in pediatric settings. VR has been shown to effectively decrease preoperative anxiety in children undergoing various medical procedures, including IV catheter replacement, blood draws, and improve their compliance with anesthesia and overall procedural experiences. Limited evidence exists regarding the impact of VR on the broader care environment, including parental anxiety and nursing satisfaction in pediatric settings.

DETAILED DESCRIPTION:
This retrospective study analyzes de-identified data from a nine-month quality improvement initiative to evaluate the impact of a custom VR intervention on pediatric preoperative anxiety, parental anxiety, and nurse satisfaction in a real clinical setting. The findings offer preliminary, practice-relevant evidence that VR can be a feasible, acceptable, and clinically meaningful non-pharmacologic tool in pediatric preoperative care, and they provide actionable insights to guide future implementation efforts and rigorous trials aimed at improving the hospital experience for children, families, and providers.

ELIGIBILITY:
Pediatric Subjects

Inclusion Criteria:

* pediatric patients who received VR intervention as part of the original QI initiative.
* pediatric patients who were eligible and received VR during the QI initiative aged 6-15 years.

Exclusion Criteria:

* Patients with developmental delays, head injuries, or seizures were excluded from the study.
* Only those pediatric patients who met the inclusion criteria and did not exhibit the specified exclusion conditions were included. Data protection and de-identification procedures were rigorously applied throughout the study

Caregivers/Parents

Inclusion Criteria:

- pediatric patients who were eligible and received VR during the QI initiative, aged 6-15 years

Exclusion Criteria:

- N/A

Nurses

Inclusion Criteria:

* nurses of pediatric patients who were eligible and received VR during the QI initiative, aged 6-15 years

Exclusion Criteria:

* N/A

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study involved pediatric patients who received VR intervention as part of the original QI initiative. Data protection and de-identification procedures were rigorously applied throughout the study
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in patient anxiety levels, as measured by heart rate | Before and after VR intervention, one visit only
  Change in patient anxiety levels, as measured by heart rate, before and after VR intervention. Baseline heart rate will be compared to the heart rate after the intervention.
Change in patient anxiety levels, as measured by blood pressure | Before and after VR intervention, one visit only
  Change in patient anxiety levels, as measured by blood pressure, before and after VR intervention. Baseline blood pressure will be compared to the blood pressure after the intervention.
Change in patient anxiety levels, as measured by distress/fear scores | Before and after VR intervention, one visit only
  Change in patient anxiety levels, as measured by distress/fear scores before and after VR intervention Baseline distress/fear scores will be compared to the distress/fear scores after the intervention. Using the Children's Fear Scale (CFS) (0-4):
  * 0 = no fear (good)
  * 4 = very high fear (bad) . Higher scores indicate worse anxiety. Anxiety levels were measured immediately before and immediately after the VR intervention).

SECONDARY OUTCOMES:
Parental anxiety levels | Before and after VR intervention, one visit only
  Change in parental anxiety levels, measured by pre- and post-intervention State-Trait Anxiety Inventory (STAI) scores. The State-Trait Anxiety Inventory (STAI) scoring involves summing the scores from the 40 items, each rated on a 4-point Likert scale, to assess state and trait anxiety. The higher the score, the higher the level of anxiety.
  1. = Not at all
  2. = Somewhat
  3. = Moderately so
  4. = Very much so
Nurse satisfaction ratings | Before and after VR intervention, one visit only
  Nurse satisfaction ratings with the VR intervention, measured via survey responses. Nurse satisfaction with the VR intervention was measured using a brief, Likert-scale survey developed for this quality improvement project.
  Survey Format: A 5-point Likert scale was used for all items:
  * 1 = Very Dissatisfied / Very Difficult (bad)
  * 2 = Dissatisfied
  * 3 = Neutral
  * 4 = Satisfied
  * 5 = Very Satisfied / Very Easy to Use (good) Higher scores indicate better satisfaction and more straightforward implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Dayanjan Wijesinghe, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No